CLINICAL TRIAL: NCT03135431
Title: Opportunistic Salpingectomy at the Time of Cesarean Delivery: A Randomized Controlled Trial of the Safety of Salpingectomy vs Tubal Ligation
Brief Title: Opportunistic Salpingectomy for Permanent Sterilization at the Time of Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vanessa Torbenson, Consultant Obstetrics and Gynecology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-000898
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salpingectomy (Experimental): Bilateral salpingectomy following cesarean delivery
  Interventions: Procedure: Bilateral Salpingectomy
- Tubal Ligation (Active Comparator): Bilateral tubal ligation following cesarean delivery via Parkland or modified Pomeroy methods.
  Interventions: Procedure: Bilateral Tubal Ligation

INTERVENTIONS:
Procedure: Bilateral Salpingectomy — Surgical removal of entire fallopian tubes
  Arms: Salpingectomy
Procedure: Bilateral Tubal Ligation — Surgical tying, cutting, or removal of a portion of the fallopian tubes
  Arms: Tubal Ligation

SUMMARY:
The purpose of this study is to compare the safety of performing a bilateral tubal ligation vs. bilateral salpingectomy, two procedures performed for permanent sterilization, at the time of cesarean delivery. The investigators want to determine if performing bilateral salpingectomy at the time of cesarean delivery poses any greater risk for blood loss, as compared to a bilateral tubal ligation.

DETAILED DESCRIPTION:
A non-inferiority, two-arm randomized controlled trial to evaluate the safety and feasibility of prophylactic salpingectomy at the time of a cesarean delivery will be conducted as an initiative to avoid a missed opportunity in the primary prevention of ovarian cancer. Once enrolled and consented, women will be randomized using a stratified block randomization algorithm according to number of prior cesarean deliveries and BMI to either salpingectomy or bilateral tubal ligation. The data collection will include preoperative CBC, time of procedure, postoperative CBC at 24 hours, standard patient demographics, procedural complications, estimated blood loss, return to the OR, length of stay, pain scores, and postoperative complications, including readmission within 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 21 years of age or older
* Desire permanent sterilization
* Scheduled for a Cesarean delivery

Exclusion Criteria:

* Body Mass Index > 50
* Emergent, 'alpha' Cesarean delivery
* Single ovary/fallopian tube complex

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-05-19 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa E Torbenson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Salpingectomy | Tubal Ligation
Started | 20 | 20
Completed | 18 | 20
Not Completed | 2 | 0
Not completed — Study Surgeon not available | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salpingectomy | Tubal Ligation | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (4.8) | 34.4 (4.1) | 33.6 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Hispanic and/or Latino | 1 | 0 | 1
  Race: White | 17 | 20 | 37
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 38
Smoking Status [Count of Participants; unit: Participants]
  Current | 5 | 3 | 8
  Former | 1 | 7 | 8
  Never | 12 | 10 | 22
Repeat Cesarean [Count of Participants; unit: Participants]
  Repeat Cesarean | 16 | 17 | 33
  First Cesarean | 2 | 3 | 5
Gestational Age [Mean (Standard Deviation); unit: weeks] | 38.0 (2.4) | 37.6 (2.6) | 37.8 (2.5)
Gravity [Median (Inter-Quartile Range); unit: Pregnancies] | 3 [2 to 5] | 4 [3 to 5] | 4 [3 to 5]
Parity [Median (Inter-Quartile Range); unit: viable pregnancies] | 1.5 [1 to 2] | 2 [1.5 to 3] | 2 [1 to 3]
Education [Count of Participants; unit: Participants]
  High school or some High School | 2 | 2 | 4
  Some College | 11 | 5 | 16
  4 year or professional degree | 5 | 12 | 17
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference Between Pre and Postoperative Hemoglobin (g/dl)
Description: Identify the mean difference in pre and postoperative hemoglobin for patients undergoing salpingectomy for sterilization vs. patients undergoing standard bilateral tubal ligation via mid-segment resection of the fallopian tube at the time of cesarean delivery.
Time Frame: At least 24 but not greater than 48 hours after surgery
Population: One patient in the Salpingectomy group is was missing post operation hemoglobin
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Salpingectomy | Tubal Ligation
Number analyzed (Participants) | 17 | 20
g/dL | 1.4 (0.7) | 1.8 (1.0)
Statistical Analysis 1: Comparison: Salpingectomy vs Tubal Ligation; Assuming that a difference of 0.5 g/dl in the drop in hemoglobin between study arms would be considered as equivalent, and assuming a common standard deviation of 1.1 based on previous studies of cesarean deliveries deliveries , the study would have 80% power to test for non-inferiority with 60 participants in each arm (120 total); Test type: Non-Inferiority — <=.5g/dl difference in the decrease in hemoglobin was considered equivalent as 1 unit of blood typically raises the hemoglobin by 1g/dl and would be a clinical significant difference; p = 0.08, t-test, 1 sided; Mean Difference (Final Values) = -.04121, 95% CI 1-sided [upper limit .0712]; Based on new data from a retrospective study preformed at Mayo Clinic sites an additional power calculation was preformed. Based on the new information, our study was well powered (84%) to assess our primary aim with 38 participants (18 salpingectomy, 20 BTL); therefore, we discontinued recruitment and completed the study with the accrued subjects

2. Secondary Outcome: Operative Time
Description: Compare mean difference in length of operative time (in minutes) to perform bilateral salpingectomy as compared to standard bilateral tubal ligation, following cesarean delivery.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: mins
Arm/Group | Salpingectomy | Tubal Ligation
Number analyzed (Participants) | 18 | 20
mins | 16.3 (5.6) | 5.1 (1.6)
Statistical Analysis 1: Comparison: Salpingectomy vs Tubal Ligation; Test type: Superiority; Mean Difference (Final Values) = -11.21, 95% CI 2-sided [-14.1 to -8.3] — Evidence to suggest salpingecotomy procedure had a longer operation time than a tubal ligation

3. Secondary Outcome: Estimated Blood Loss
Description: Identify mean difference in estimated total blood loss as a result of standard bilateral tubal ligation surgical procedure and bilateral salpingectomy procedure, following cesarean delivery.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Salpingectomy | Tubal Ligation
Number analyzed (Participants) | 18 | 20
mL | 842 (84.5) | 833 (105.5)
Statistical Analysis 1: Comparison: Salpingectomy vs Tubal Ligation; Analysis preformed as categorical and categorical variable. Both analyzes had the same conclusion; Test type: Superiority; p = 0.77, t-test, 2 sided; Mean Difference (Net) = -9.17, 95% CI 2-sided [-72.5 to 54.17]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on participants six weeks from the date of cesarean delivery.
Description: Definition also included the following statement: "problems/events that in the opinion of the PI may have adversely affected the rights, safety, or welfare of the subjects or others, or substantially compromised the research data."
Groups:
- Salpingectomy: Bilateral salpingectomy (surgical removal or entire fallopian tubes) following cesarean delivery
- Tubal Ligation: Bilateral tubal ligation (surgical tying, cutting, or removal of a portion of the fallopian tubes)following cesarean delivery via Parkland or modified Pomeroy methods.
Arm/Group | Salpingectomy | Tubal Ligation
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/18 | 0/20
Other Adverse Events (participants affected / at risk) | 1/18 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salpingectomy (N=18) | Tubal Ligation (N=20)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — Grade 1
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 2
Uterine hemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) — Grade 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salpingectomy (N=18) | Tubal Ligation (N=20)
Other, post-operative pain score above goal (Surgical and medical procedures) | 0 (0) | 1 (1) — Grade 1
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Grade 2
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03135431/Prot_SAP_ICF_000.pdf